CLINICAL TRIAL: NCT03286504
Title: FANMI: Community Cohort Care for HIV-Infected Adolescent Girls in Haiti
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Haitian Group for the Study of Kaposi's Sarcoma and Opportunistic (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1504016098; R01HD091935 (NIH)
Record Dates: First submitted 2017-09-13; First posted 2017-09-18 (Actual); Results first posted 2023-06-02 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: HIV

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard-of-care (No Intervention): Adolescents randomized to the standard arm will receive monthly HIV care in the GHESKIO Adolescent Clinic. Clinical care is provided in an individual exam room by a nurse. The patient is sequentially referred to the laboratory, social worker, and pharmacy for medication refills. A typical visit, including wait time, lasts 3 hours.
- FANMI - Cohort Care (Experimental): Adolescents randomized to FANMI will receive all monthly HIV care in the community room of the Prince Albert School in Village of God. Adolescents will be grouped in cohorts of 5-10 peers. The entire visit will take ~ 2 hours.
  Interventions: Behavioral: FANMI - Cohort Care

INTERVENTIONS:
Behavioral: FANMI - Cohort Care — FANMI includes receiving integrated clinical care, group counseling, and social activities in a single session by the same provider to simplify care and strengthen relationships between peers and providers. FANMI groups consist of 5-10 adolescents meeting once per month.
  Arms: FANMI - Cohort Care

SUMMARY:
The investigators will conduct a randomized controlled trial of Group Care in the GHESKIO Community Center versus Individual Care in the GHESKIO Adolescent Clinic for 160 HIV-infected adolescent girls age 16-23 years in Haiti (80 adolescents per arm). Group Care includes receiving integrated clinical and social support services in groups of 5-8 adolescents at a monthly visit. The primary outcome is retention in HIV care at 12 months after randomization.

DETAILED DESCRIPTION:
The investigators will conduct a randomized controlled trial of Group Care in the GHESKIO Community Center versus Individual Care in the GHESKIO Adolescent Clinic for 160 HIV-infected adolescent girls age 16-23 years in Haiti (80 per arm). Adolescents randomized to Group Care will receive HIV services including integrated clinical and social support care in groups of 5-10. Adolescents randomized to Individual Care will continue to receive individual care at the GHESKIO Adolescent Clinic, which is the current standard of care (described below). If a subject declines to participate in the study they will continue to receive standard HIV care. Participants will be randomized to either Group Care or Individual Care in a 1:1 ratio using a computer generated random assignment.

Individual Care (standard of care): Adolescents randomized to Individual Care will receive care in the GHESKIO Adolescent Clinic which cares for both males and females age 13-23 years. The Adolescent Clinic waiting room has a television showing educational videos. After seeing a triage peer counselor and having their vital signs taken, participants see a nurse practitioner (NP) one-on-one in a private room for a 10-15 minute clinic visit. The NP may also provide family support counseling including family visits per clinical judgment. Each NP sees approximately 20 HIV-infected adolescents per day. The adolescent then returns to the HIV positive peer counselor, who provides one-on-one counseling for 30 minutes on topics chosen by the adolescent and the counselor. Each counselor sees ~10 adolescents per day.

Group Care (intervention): Adolescent girls randomized to Group Care will join a group within one week of study enrollment and receive care in the GHESKIO Community Center. The investigators estimate that it will take 4-6 weeks to constitute a full group of 5-10. During this enrollment phase, groups will meet weekly, adding new participants each week. The participants will then meet monthly with an NP and a HIV positive peer counselor. Each monthly group session will last ~2 hours. This is comparable to the time it takes for a patient to pass through the Adolescent HIV Clinic. It will start with a 30 minute unstructured discussion. This time is intentionally unstructured and responds to our previous research finding that adolescents want to talk about topics of their choosing with their peers. This will be followed by a 45 minute group counseling session following a structured curriculum, addressing topics such as social isolation, stigma, family support, sexual risk behavior, life goals, medication adherence, job skills, and transitions. This is followed by a 30 minute social activity led by two rotating group leaders who are elected by their peers. Social activities include crafts, playing cards, and charades. Participants will be seen one by one by the NP for ~10-15 minutes in a screened in clinical area during the unstructured discussion and the social activity. All HIV clinical services, including provision of antiretroviral therapy (ART) medications, CD4 T cell monitoring, screening for symptoms and OI, medication adherence monitoring, family planning, and general primary care will be provided by the NP. Girls who become eligible for ART will be provided with individual counseling and promptly initiated on ART by the NP. The primary hypothesis is that Group Care will improve retention at 12 months compared with standard Individual Care. The study has > 90% power to detect a difference in retention from 60% to 85%. Participants in both study arms will complete a questionnaire with a research nurse at enrollment, 6, and 12 months collecting data on HIV knowledge, HIV-related stigma, HIV disclosure, social and family support, depression and alcohol use, problem solving skills, and food insecurity.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 16-23 years
* ART naive, initiated ART in the past 3 months, or defaulted from care for 3 months or more
* Participant knowledge of HIV-infection
* Willing to receive care at the clinic or in the community
* Willing to provide consent (age 18 -23 years) or assent with parental/guardian consent (16-17 years)

Exclusion Criteria:

* Pregnancy at the time of enrollment
* A severe HIV/AIDS illness requiring hospitalization or intensive medical follow-up
* Based on the primary clinician's judgement that the adolescent is at a developmental stage not suited for study participation

Ages: 16 Years to 23 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — The HIV epidemic in Haiti disproportionally affects adolescent girls age 16-23. Our study involves recruitment and enrollment of adolescent girls to determine if our intervention is effective in retaining HIV-infected adolescent girls in Haiti.
Enrollment: 120 (Actual)
Dates: Start 2018-05-25 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2023-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Fitzgerald, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- GHESKIO, Port-au-Prince, Haiti

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared once the trial is complete

REFERENCES:
- [Derived] Seo G, Joseph JMB, Confident N, Jean E, Louis B, Bell T, Riche RC, Belizaire ME, Rouzier V, Apollon A, Reif L, Rivera V, Abrams E, Bang H, Schackman B, Fitzgerald D, Pape JW, McNairy ML. The FANMI ("my FAMILY" in Creole) study to evaluate community-based cohort care for adolescent and young women living with HIV in Haiti: protocol for a randomized controlled trial. BMC Public Health. 2019 Dec 30;19(1):1749. doi: 10.1186/s12889-019-8065-6. PMID 31888569

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard-of-care | FANMI - Cohort Care
Started | 60 | 60
Completed | 41 | 44
Not Completed | 19 | 16
Not completed — Lost to Follow-up | 19 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard-of-care | FANMI - Cohort Care | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 10 | 16
  Between 18 and 65 years | 54 | 50 | 104
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 60 | 120
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 60 | 60 | 120
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 60 | 60 | 120
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: 12 Month Retention
Description: Retention in care at 12 months will be measured. 12 month retention is defined as being alive at 12 months and having a care visit between 9 and 15 months after enrollment.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard-of-care | FANMI - Cohort Care
Number analyzed (Participants) | 60 | 60
Participants | 41 | 44
Statistical Analysis 1: Comparison: Standard-of-care vs FANMI - Cohort Care; Test type: Superiority; p = 0.55, Chi-squared; proportion difference = 0.05, 95% CI 2-sided [-0.112 to 0.212] — Direction of proportion difference = FANMI arm minus Standard of Care arm

2. Secondary Outcome: 12 Month Viral Suppression
Description: Viral suppression at 12 months will be measured. Suppressed viral load will be defined as a binary outcome based upon the WHO definition of viral suppression as a plasma HIV-1 RNA level <1000 copies/µl.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard-of-care | FANMI - Cohort Care
Number analyzed (Participants) | 60 | 60
Participants | 26 | 28
Statistical Analysis 1: Comparison: Standard-of-care vs FANMI - Cohort Care; Test type: Superiority; p = 0.71, Chi-squared; proportion difference = 0.033, 95% CI 2-sided [-0.145 to 0.211] — Direction of proportion difference = FANMI arm minus Standard of Care arm

3. Secondary Outcome: Time to Antiretroviral Therapy (ART) Initiation
Description: Time to ART initiation is the number of calendar days from date of HIV diagnosis to date of ART initiation.
Time Frame: 12 months
Population: Participants analyzed were only those who were ART-naïve at study enrollment.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Standard-of-care | FANMI - Cohort Care
Number analyzed (Participants) | 34 | 33
days | 0 [0 to 0] | 0 [0 to 0]

4. Secondary Outcome: Optimal Antiretroviral Therapy (ART) Adherence
Description: ART adherence will be measured by self-report using two questions: 1) number of pills missed in the past 4 days and 2) forgot to take pills last weekend. A response of no missed pills in the past 4 days and did not forget to take pills last weekend is defined as 'optimal' adherence. All other responses are defined as 'sub-optimal' adherence.
Time Frame: 12 months
Population: There were 18 participants in the SOC arm and 22 participants in the FANMI arm who chose not to respond to the ART adherence assessment and were not included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard-of-care | FANMI - Cohort Care
Number analyzed (Participants) | 42 | 38
Participants | 22 | 18
Statistical Analysis 1: Comparison: Standard-of-care vs FANMI - Cohort Care; Test type: Superiority; p = 0.65, Chi-squared; proportion difference = -0.05, 95% CI 2-sided [-0.269 to 0.169] — Direction of proportion difference = FANMI arm minus Standard of Care arm

5. Secondary Outcome: Sexual Risk Behavior
Description: Sexual risk behavior will be measured by regular condom use among those who are sexually active. Regular condom use is defined as a response of 'often' or 'always' when asked about condom use during sexual intercourse.
Time Frame: 12 months
Population: There were 21 participants in the SOC arm and 26 subjects in the FANMI arm that did not receive STI testing and were excluded from this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard-of-care | FANMI - Cohort Care
Number analyzed (Participants) | 39 | 34
Participants | 21 | 26
Statistical Analysis 1: Comparison: Standard-of-care vs FANMI - Cohort Care; Test type: Superiority; p = 0.04, Chi-squared; proportion difference = 0.226, 95% CI 2-sided [0.015 to 0.438] — Direction of proportion difference = FANMI arm minus Standard of Care arm

6. Secondary Outcome: Number of Sexually Transmitted Infections
Description: Sexually Transmitted Infections will include syphilis, diagnosed using a serum RPR (HUMAN) followed by a treponemal test if positive (Bioline Standard Diagnostics), chlamydia and gonorrhea, diagnosed by the urine GeneXpert GT/NG assay.
Time Frame: 12 months
Population: There were 14 participants in the SOC arm and 13 subjects in the FANMI arm that did not receive STI testing and were excluded from this analysis.
Measure: Number; unit: incident STI diagnoses
Arm/Group | Standard-of-care | FANMI - Cohort Care
Number analyzed (Participants) | 46 | 47
incident STI diagnoses | 10 | 20
Statistical Analysis 1: Comparison: Standard-of-care vs FANMI - Cohort Care; Test type: Superiority; p = 0.03, Chi-squared; proportion difference = 0.208, 95% CI 2-sided [0.023 to 0.393] — Direction of proportion difference = FANMI arm minus Standard of Care arm

7. Secondary Outcome: Acceptability
Description: FANMI Acceptability will be assessed using qualitative interviews conducted at 6 and 12 months after study enrollment with a subset of 30 FANMI participants and clinic providers (nurses and peer educators). A trained qualitative research assistant will interview adolescents to explore attitudes about the FANMI intervention, specifically as it relates to social isolation, stigma, and family rejection, self-esteem and clinic-level factors.
Time Frame: 12 months
Population: Data for this outcome was not collected.
Arm/Group | Standard-of-care | FANMI - Cohort Care
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Healthcare Utilization
Description: Healthcare utilization will be measured. Healthcare utilization will be measured as a composite of attendance at HIV care visits, laboratory services, and use of other specialist services at study sites and use of health services at non-study sites such as hospitalizations or visits to other medical specialists.
Time Frame: 12 months
Population: Data not collected.
Arm/Group | Standard-of-care | FANMI - Cohort Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Standard-of-care | FANMI - Cohort Care
All-Cause Mortality (participants affected / at risk) | 0/60 | 1/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-12): https://cdn.clinicaltrials.gov/large-docs/04/NCT03286504/Prot_SAP_000.pdf